CLINICAL TRIAL: NCT02567578
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Dose-finding Phase 2 Trial to Evaluate the Efficacy and Safety of YH12852 in Patients With Functional Dyspepsia
Brief Title: A Trial to Evaluate the Efficacy and Safety of YH12852 in Patients With Functional Dyspepsia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Technology transfer
Sponsor: Yuhan Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: YH12852-201
Record Dates: First submitted 2015-10-01; First posted 2015-10-05 (Estimated); Last update posted 2022-01-13 (Actual); Status verified 2021-12

CONDITIONS: Functional Dyspepsia
MeSH Terms: interventions — YH12852

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- YH12852 0.1 mg (Experimental): twice daily for 4 weeks
  Interventions: Drug: YH12852 0.1 mg
- YH12852 0.25 mg (Experimental): twice daily for 4 weeks
  Interventions: Drug: YH12852 0.25 mg
- YH12852 0.5 mg (Experimental): twice daily for 4 weeks
  Interventions: Drug: YH12852 0.5 mg
- Placebo (Placebo Comparator): twice daily for 4 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: YH12852 0.1 mg
  Arms: YH12852 0.1 mg
Drug: YH12852 0.25 mg
  Arms: YH12852 0.25 mg
Drug: YH12852 0.5 mg
  Arms: YH12852 0.5 mg
Drug: Placebo
  Arms: Placebo

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled dose-finding phase 2 trial to evaluate the efficacy and safety of YH12852 in patients with functional dyspepsia.

DETAILED DESCRIPTION:
Eligible subjects will be randomized into one of 4 groups; YH12852 0.1 mg, 0.25 mg, 0.5 mg, or placebo at the same ratio and will be administered investigational products orally, twice daily for 4 weeks and followed up for 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be willing and able to provide written informed consent.
2. BMI of < 35 kg/m2
3. Patients experiencing one or more of functional dyspepsia symptoms beginning at least 6 months prior according to Rome III criteria, with the symptom(s) evident over the last 3 months at the time of screening
4. Patients with no evidence of organic lesions based on upper GI endoscopy, which could be the cause of dyspeptic symptoms
5. Women of childbearing potential (WOCBP) must have a negative pregnancy test result at the screening visit and use an adequate method of contraception to avoid pregnancy throughout the study

Exclusion Criteria:

1. Women who are pregnant or breastfeeding.
2. Women with a positive pregnancy test result on enrollment or prior to investigational product administration.
3. Subjects with a history of surgery that could affect gastrointestinal motility
4. Subjects with inflammatory bowel disease
5. Clinically significant chronic infection (eg. AIDS, etc), or significant medical or psychiatric illness.
6. Serious cardiovascular disease (including QT prolongation defined as QTc interval ≥ 450msec) or respiratory disease
7. History of alcohol or drug abuse within the previous one year.
8. Subjects with mental illness (e.g. schizophrenia, dementia etc) that may render the inability to complete the study
9. Physical and Laboratory Test Findings
10. Administration of any other investigational product or participation in other clinical trials within 3 months prior to randomization.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2015-10; Primary Completion 2017-03-16 (Actual); Study Completion 2017-03-16 (Actual)

PRIMARY OUTCOMES:
Ratio of OTE (Overall Treatment Efficacy) responders | 4 weeks

SECONDARY OUTCOMES:
Ratio of OSS responders | 4 weeks
Elimination rate for 8 functional dyspepsia symptoms | 4 weeks
Change from basline in NDI QoL score | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Poong Lyul Lee, MD, Ph.D, Principal Investigator — Samsung seoul hospital
Locations (1):
- Samsung seoul hospital, Seoul, South Korea